CLINICAL TRIAL: NCT04452552
Title: Effect of Ultrasound Cavitation Versus Radiofrequency on Abdominal Fat Thickness in Postnatal Women
Brief Title: Ultrasound Cavitation Versus Radiofrequency on Abdominal Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Yasmin Mohamed Assim (Unknown)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 98
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Healthy Diet
Keywords: Ultra-sound cavitation; Radiofrequency; fat thickness
MeSH Terms: interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Fifty overweight primipara women at 6 months postnatally aged from 20-35 years, BMI (25-29.9) kg/m2 and have waist hip ratio (WHR) > 0.8. They were assigned randomly into 2 equal groups: Group (A) received ultra-sound cavitation40 KHz applied for 30 min, once time weekly for 8 weeks. Group (B) received radiofrequency multi-polar 5MHZ applied for 30 min, once time weekly for 8 weeks. Both groups received the same diet program throughout the treatment period. All females in both groups were assessed through weight scale for body weight, tape measurement for waist/hip ratio and ultra-sonography for fat thickness of abdominal region before and after treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: An independent person randomly assigned to all participated subjects to either group (A) or group (B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultra-sound cavitation (Experimental): cavitation40 KHz applied for 30 min, once time weekly for 8 weeks.
  Interventions: Other: healthy diet
- radiofrequency (Experimental): radiofrequency multi-polar 5MHZ applied for 30 min, once time weekly for 8 weeks
  Interventions: Other: healthy diet

INTERVENTIONS:
Other: healthy diet — balanced diet program which ranged from 1600 kcal to 2000 kcal/day, which was calculated in an individual basis for each woman according to her basal metabolic rate (BMR) for 8 weeks

SUMMARY:
Overweight and obesity is prevalent among women of reproductive age (25-34 years) with 42% having a BMI > 25 kg/m2. Weight gain increases the risk of developing diabetes and cardiovascular disease. The amount of weight regain postpartum can shift women from the healthy weight category into the overweight or obese BMI categories. Purpose: This study was conducted to compare the effectiveness of ultra-sound Cavitation versus radiofrequency on abdominal fat thickness on postnatal women

DETAILED DESCRIPTION:
Fifty overweight primipara women at 6 months postnatally aged from 20-35 years, BMI (25-29.9) kg/m2 and have waist hip ratio (WHR) > 0.8. They were assigned randomly into 2 equal groups: Group (A) received ultra-sound cavitation40 KHz applied for 30 min, once time weekly for 8 weeks. Group (B) received radiofrequency multi-polar 5MHZ applied for 30 min, once time weekly for 8 weeks. Both groups received the same diet program throughout the treatment period. All females in both groups were assessed through weight scale for body weight, tape measurement for waist/hip ratio and ultra-sonography for fat thickness of abdominal region before and after treatment

ELIGIBILITY:
Inclusion Criteria:

* Their age were ranged from 20 to 35 years
* their body mass index BMI 25-29.9 kg/m2
* their waist hip ratio (WHR) > 0.8.

Exclusion Criteria:

* heart disease
* high cholesterol
* liver
* kidney diseases

Ages: 25 Years to 35 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01-24 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
BMI calculation | 8 weeks
  The woman's BMI had calculated from measured weight & height for each woman in both groups (A&B) before beginning of the study and weight only had measured after 8 weeks of treatment sessions to according to the following equation: BMI=weight (Kg) /height (m2)

SECONDARY OUTCOMES:
Waist to hip ratio Measurement | 8 weeks
  WHR was calculated by dividing WC on HC. Both measurements were taken for all women in all groups (A & B) before starting the study and after 8 weeks of treatment sessions (end of study). All measurements were with the women in standing position. Skin of the anterior abdominal wall was cleaned while the woman in hip circumference worn light clothes and sometimes measurements repeated twice for more accurate. That measured WC, HC to measure (WHR) calculated by dividing the measurement of the waist by the measurement of the hips.
  WHR= (waist circumference / hip circumference)

CONTACTS AND LOCATIONS:
Overall Officials: ghada eb elrefaye, professor, Principal Investigator — Cairo University
Locations (1):
- Ghada Elrefaye, Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided